CLINICAL TRIAL: NCT00520507
Title: An Investigation of the Sleep Architecture and Consequent Cognitive Changes in Olanzapine-Treated Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Prinicpal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSIY-263-07
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorder; Depression; Depressive Disorder
Keywords: Depression; Bipolar Disorder; Major
MeSH Terms: conditions — Bipolar Disorder; Depression; Depressive Disorder | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Olanzapine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — Olanzapine will be taken once daily at 6pm for 1 month. Dosing will be titrated up to 5mg and then changed as clinically indicated.
  Arms: 1
Drug: Placebo — An inactive form of the treatment will be taken once daily at 6pm for 1 month.
  Arms: 2

SUMMARY:
OBJECTIVES:

Primary Objective:

To assess the objective (polysomnographic) changes in sleep quality before and after introduction of olanzapine in treatment of patients with depression.

Secondary Objectives:

To assess the subjective changes in sleep quality parameters before and at different stages after introduction of olanzapine in treatment, longitudinally, and to correlate these changes with measures of illness severity and changes in cognition.

STUDY DESIGN:

Prospective, double blind, randomized polysomnographic (PSG) study of patients before and after treatment with olanzapine.

PSG recordings will be done three times throughout the study: before starting olanzapine augmentation (baseline), at day 3 to 5 (acute) and day 28 to 31 (chronic). PSG will be completed at patients' homes with a portable PSG. Psychiatric scales, subjective sleep quality scales, and cognition measurements will be completed at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of major depressive disorder or bipolar disorder type 1, 2 or NOS by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
2. Current depressive episode with a HAMD-17 of > 15
3. Males or females over age18 years (yrs)
4. Inpatients or outpatients
5. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
6. Able to understand and comply with the requirements of the study
7. Provision of written informed consent

Exclusion Criteria:

1. Current manic, hypomanic or mixed episode, with YMRS > 12
2. Current or past diagnosis of schizophrenia and dementia
3. Pregnant women, or women in childbearing age, not willing to use appropriate contraception or women currently nursing
4. Patient on any other antipsychotic medication
5. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
6. Known intolerance or lack of response to olanzapine, as judged by the investigator
7. Benzodiazepines and all other sleep-aids must be discontinued prior to participation in the study if they have not been at a stable dosage for the 4 weeks previous to entry into the study
8. No change to the current medication regime (excluding discontinuation of sleep aids and antipsychotic medications) is allowed 4 weeks prior to the first PSG reading
9. Administration of a depot antipsychotic injection within two dosing interval (for the depot) before randomization
10. Substance or alcohol dependence at enrolment or in the last three months (except for caffeine or nicotine dependence), as defined by DSM-IV criteria
11. Serious, unstable or inadequately treated medical illness as judged by the investigator
12. History of epilepsy or uncontrolled seizures
13. Involvement in the planning and conduct of the study
14. Previous enrolment in the present study
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Sleep quality as measured by overnight PSG, defined as the change in time spent in slow wave sleep. | 3 days after baseline and 1 month after baseline

SECONDARY OUTCOMES:
Sleep measures: time in bed, total sleep time, sleep period time, percentage of sleep stages (stage 1, stage 2, slow wave sleep, REM sleep) of sleep period time, sleep latency to stage 1 and 2, REM latency, number of awakenings. | measure taken at baseline, 3 days after baseline, and 1 month after baseline
Respiratory events (during PSG): obstructive sleep apneas, mixed apneas, central apneas, total apneas, obstructive hypopneas, mixed hypopneas, central hypopneas, total hypopneas, and apneas + hypopneas (AHI), oxygen saturation, and heart rate. | Baseline, 3 days and 1 month after baseline
Subjective sleep experience: visual analogue scale, sleep diary, Epworth Sleep Scale and Pittsburgh Sleep Quality Index. | Baseline, 3 days and 1 month after baseline
Changes in weight and blood glucose will be monitored. | At baseline and 1 month
Cognition: CANTAB scores | Baseline, 3 days and 1 month after baseline
Illness severity: HDRS-17, MADRS, CGI and HamA | Baseline, 3 days and 1 month after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, M.D., Principal Investigator — Queen's University, Department of Psychiatry
Locations (1):
- Queen's University, Providence Care-Mental Health Services, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Lazowski LK, Townsend B, Hawken ER, Jokic R, du Toit R, Milev R. Sleep architecture and cognitive changes in olanzapine-treated patients with depression: a double blind randomized placebo controlled trial. BMC Psychiatry. 2014 Jul 17;14:202. doi: 10.1186/1471-244X-14-202. PMID 25030264